CLINICAL TRIAL: NCT06351930
Title: Efficacy of Cognitive Behaviour Therapy for Insomnia (CBT-I) in Adolescents With Attention Deficit Hyperactivity Disorder (ADHD): A Randomized Controlled Trial
Brief Title: CBT for Insomnia in Adolescents With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Kwai Chung Hospital (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA210473
Record Dates: First submitted 2024-04-01; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Insomnia; ADHD
Keywords: Insomnia; ADHD; Adolescents; Youth; CBT-I
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: A randomised, assessor-blind, parallel group controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive behaviour therapy for insomnia (CBT-I) + usual care (UC) group (Experimental): The intervention for the CBT-I + UC group will involve five weekly 50-minute individual, face-to-face sessions of CBT-I. The treatment components aim to address the behavioural, cognitive and physiological perpetuating factor of insomnia whilst considering the clinical context of ADHD and include: psycho-education about ADHD, sleep, circadian rhythm and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention.
  Interventions: Behavioral: CBT-I + UC group
- UC group (No Intervention): Participants will continue their usual clinical follow-up and receive standard treatment at the clinic.

INTERVENTIONS:
Behavioral: CBT-I + UC group — Refer to the arm description
  Arms: cognitive behaviour therapy for insomnia (CBT-I) + usual care (UC) group

SUMMARY:
Insomnia and attention deficit hyperactivity disorder (ADHD) are highly comorbid conditions with an intricate, bidirectional relationship. In particular, insomnia and ADHD often co-occur, with 22.9-34.6% of adolescents with insomnia having clinically significant ADHD, and 22-33.5% of adolescents with ADHD experiencing comorbid insomnia symptoms. Insomnia is not only associated with increased ADHD severity, but also linked to an increased risk for other mental health problems and poorer treatment response in young people with ADHD. Behavioural sleep interventions have shown promise in improving sleep in young children with comorbid ADHD and insomnia. Nonetheless, when treating adolescent insomnia, especially those with ADHD, there is a need to consider the unique sleep and circadian features as well as psychosocial factors associated with not only ADHD but also adolescence, a challenging developmental stage. To date, there is a paucity of research to test the efficacy of cognitive behavioural therapy for insomnia (CBT-I) in adolescents with comorbid ADHD and insomnia. To address the limitations in the existing literature, this study aims to conduct a randomised controlled trial (RCT) to examine the effects of CBT-I relative to a usual care (UC) condition in adolescents with ADHD, on improving sleep and ADHD symptoms, and other clinical and daytime symptoms as well as overall functional improvement.

DETAILED DESCRIPTION:
An assessor-blind, parallel-group, randomised controlled trial will be conducted in adolescents with comorbid ADHD and insomnia. Eligible participants will be randomised to either CBT-I + UC or UC condition. Assessments will be conducted at baseline (T1), one-week post-treatment (T4), and post-treatment 3-month (T5). In addition, participants in both conditions will complete the Insomnia Severity Index (ISI) at T2 (week 2) and T3 (week 4) during the intervention. A random sample of 15 participants per group will be assessed for sleep objectively using actigraphy for 7 consecutive days at baseline (T1) and one-week post-treatment (T4). Participants in the control group will be offered CBT-I after post-treatment 3-month follow-up. During the study period, all the participants will continue their regular clinical follow-ups with their attending psychiatrist for the prescription of psychotropic medication(s), if needed, for managing their ADHD and mental health condition. Prescription of any psychotropic medications of each participant during the trial will be reviewed and documented at baseline and at each follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Cantonese-speaking adolescent aged 12-18 years old;
2. A diagnosis of ADHD as confirmed by the Diagnostic Interview Schedule for Children-version-IV (DISC-IV);
3. Having a DSM-5 diagnosis of insomnia disorder and with a score on Insomnia Severity Index (ISI) ≥ 9 (suggested cut-off for adolescents);
4. Written informed consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18);
5. Being able to comply with the study protocol;
6. Those who are not on ADHD medication or have been stabilized on psychostimulant or nonstimulant ADHD medications (maintaining the optimal medication dosage for at least 6 months).

Exclusion Criteria:

1. A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, autism spectrum disorder, organic mental disorders, or intellectual disabilities;
2. Having a prominent medical condition known to interfere with sleep continuity and quality (e.g., severe eczema, gastro-oesophageal reflux disease);
3. Having a clinically diagnosed sleep disorder that may potentially contribute to a disruption in sleep continuity and quality, such as narcolepsy, sleep-disordered breathing, and restless leg syndrome;
4. Concurrent, regular use of psychotropic medications(s) known to affect sleep continuity and quality (e.g., hypnotics, steroids), except for the use of psychostimulant medication for ADHD;
5. Receiving ongoing psychological treatment for sleep problems;
6. With hearing or speech deficit;
7. In the opinion of the research clinician, having a clinically significant suicidality (e.g., with suicidal ideation with a plan or a suicide attempt in the recent one month), and/or endorsing "nearly everyday" for item 9 (suicidal thoughts) in the Patient Health Questionnaire - 9 (PHQ-9).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Symptoms | Baseline, week 2&4 of the intervention, one-week post-treatment and post-treatment 3 month.
  Insomnia symptoms measured by Insomnia Severity Index (ISI). ISI is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.

SECONDARY OUTCOMES:
Change in ADHD Symptoms (Self-report) | Baseline, one-week post-treatment and post-treatment 3 month
  The Adult ADHD Self-Report Scale (ASRS) v1.1 Symptom Checklist is an 18-item self-administered questionnaire to screen for ADHD symptoms in both community surveys and clinical settings based on criteria of the DSM-IV-TR. The questionnaire asks participants to rate how often a symptom of inattention or hyperactivity has occurred during the past 6 months using a scale from 0 (never) to 4 (very often). The total score on this scale can range from 0 to 72, with higher scores indicating more ADHD symptomology.
Change in Internalising and Externalising Symptoms (Parent-rated) | Baseline, one-week post-treatment and post-treatment 3 month
  The Strengths and Difficulties Questionnaire (SDQ) - parent report is a widely used and validated screening questionnaire to measure emotional and behavioural problems in adolescents. It consists of 25 items covering five subscales relating to emotional problems, peer problems, conduct problems, hyperactivity, and prosocial behaviour. A higher score of the scales indicates a higher severity of the problem, except for prosocial behaviour scale.
Change in depressive symptoms (Self-report) | Baseline, one-week post-treatment and post-treatment 3 month
  Patient Health Questionnaire - 9 (PHQ9) consists of nine items to assess the frequency of depressive symptoms in the past 2 weeks. Higher scores suggest more severe depressive symptoms.
Change in anxiety symptoms (Self-report) | Baseline, one-week post-treatment and post-treatment 3 month
  Generalized Anxiety Disorder 7-item scale (GAD-7) is a self-report measure of generalised anxiety symptoms in the past 2 weeks. Higher scores suggest more severe anxiety symptoms.
Change in Sleep Diary Measure - Time in Bed (TIB) | Baseline, one-week post-treatment and post-treatment 3 month
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours
Change in Sleep Diary Measure - Total Sleep Time (TST) | Baseline, one-week post-treatment and post-treatment 3 month
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours
Change in Sleep Diary Measure - Sleep Onset Latency (SOL) | Baseline, one-week post-treatment and post-treatment 3 month
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (SOL) in mins
Change in Sleep Diary Measure - Wake After Sleep Onset (WASO) | Baseline, one-week post-treatment and post-treatment 3 month
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (WASO) in mins
Change in Sleep Diary Measure - Sleep Efficiency (SE) | Baseline, one-week post-treatment and post-treatment 3 month
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change in Objective Sleep Measures - Time in Bed (TIB) | Baseline and one-week post-treatment
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: time in bed (TIB) in hours. A subset of sample will complete actigraphic assessment.
Change in Objective Sleep Measures - Total Sleep Time (TST) | Baseline and one-week post-treatment
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: total sleep time (TST) in hours. A subset of sample will complete actigraphic assessment.
Change in Objective Sleep Measures - Sleep Onset Latency (SOL) | Baseline and one-week post-treatment
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep onset latency (SOL) in mins. A subset of sample will complete actigraphic assessment.
Change in Objective Sleep Measures - Wake After Sleep Onset (WASO) | Baseline and one-week post-treatment
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: wake after sleep onset (WASO) in mins. A subset of sample will complete actigraphic assessment.
Change in Objective Sleep Measures - Sleep Efficiency (SE) | Baseline and one-week post-treatment
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %. A subset of sample will complete actigraphic assessment.
Change in Individual Beliefs and Attitude about Sleep | Baseline, one-week post-treatment and post-treatment 3 month
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 16-item self-rated scale measuring the respondent's sleep-related beliefs, more specifically, their expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. A total score is calculated by averaging score of all items, possibly scored 0 to 10, with a higher score indicating more dysfunctional beliefs and attitudes about sleep.
Change in Adolescent Sleep Hygiene | Baseline, one-week post-treatment and post-treatment 3 month
  The Revised Adolescents Sleep Hygiene Scale (ASHSr) is used to measure adolescent sleep hygiene. It comprises 33 self-report items, categorizing into six subscales: physiological, sleep environment, cognitive/emotional, sleep stability, daytime sleep, and behavioral arousal. Adolescents rate the frequency of their sleep-related behaviors over the past month using a 6-point scale, where 1 corresponds to "always" and 6 to "never." Subscale scores are computed using means, and these scores range from 1 to 6. Higher scores on the subscales indicate better sleep hygiene.
Change in Quality of Life | Baseline, one-week post-treatment and post-treatment 3 month
  KIDSCREEN-27 is a 27-item self-rated scale measuring health related quality of life measure for children and adolescents. There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Child and adolescent outpatient psychiatric clinic of Kwai Chung Hospital, Hong Kong
  - Sleep Research Clinic and Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No